CLINICAL TRIAL: NCT05065554
Title: Phase II Study on Acalabrutinib and Anti-CD20 Antibody in Patients With Predominantly Demyelinating Neuropathy With or Without Anti-MAG
Brief Title: ACALA-R In Predominantly Demyelinating IgM Mediated Neuropathy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shayna Sarosiek, MD (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Shayna Sarosiek, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-439
Record Dates: First submitted 2021-09-20; First posted 2021-10-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: IgM MGUS; Waldenstrom Macroglobulinemia; Neuropathy;Peripheral
Keywords: IgM MGUS; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Neuritis | interventions — acalabrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ACALABRUTINIB + RITUXIMAB/BIOSIMILAR (Experimental): Acalabrutinib and rituximab (or biosimilar) with be contained in the treatment regimen.
  Acalabrutinib will be administered twice daily, with 28 consecutive days defined as a treatment cycle. Acalabrutinib will be administered for 48 cycles or until disease progression or unacceptable toxicity.
  Rituximab will be administered on Days 1, 8, 15, and 22 of Cycles 1 and 4. Participants will have study visits every cycle for cycles 1-6, then every 3 cycles, with the next visit at Cycle 9, then C12, C15, etc.
  Participants will continue acalabrutinib until disease progression or intolerable adverse effect develops. They will be followed for up to 2 years after completion of 48 cycles of treatment or until death
  Interventions: Drug: Acalabrutinib; Drug: Rituximab

INTERVENTIONS:
Drug: Acalabrutinib — Dose per protocol, oral twice daily per cycle
  Other Names: Calquence
Drug: Rituximab — Premedications (including acetaminophen, an antihistamine, and a steroid) will be given per institutional guideline Dosage determined per protocol and cycle timepoint, Route IV or SQ per protocol and cycle timepoint, schedule per protocol and cycle timepoint
  Other Names: Rituxan

SUMMARY:
In this research study, is combining a new treatment acalabrutinib with a standard treatment, rituximab or other CD20 antibody, to determine whether this combination is safe and effective for participants with Immunoglobulin (Ig) M monoclonal gammopathy of undetermined significance ( IgM MGUS) or Waldenström macroglobulinemia WM related neuropathies.

The names of the study drugs involved in this study are/is:

* Acalabrutinib
* Rituximab or similar CD20 antibody

DETAILED DESCRIPTION:
This research study involves an experimental drug combination of a targeted therapy and a CD20 antibody.

The names of the study drugs involved in this study are/is:

* Acalabrutinib
* Rituximab or similar CD20 antibody

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

The study treatment for up to 4 years and will be followed for 2 years after completion of study treatment.

It is expected that about 33 people will take part in this research study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved acalabrutinib for this specific disease but it has been approved for other uses.

The U.S. Food and Drug Administration (FDA) has not approved rituximab or similar CD20 antibody for this specific disease but it has been approved for other uses.

* Acalabrutinib is a targeted therapy that blocks a type of protein called Bruton Tyrosine Kinase (BTK) that helps cells live and grow. By blocking BTK, acalabrutinib may kill abnormal cells or stop them from growing. It has been FDA approved for mantle cell lymphoma (MCL).
* Rituximab, or biosimilar, is a type of therapy called an antibody that attacks CD20, a protein found on B-cells. Rituximab is approved by the FDA for treating non-Hodgkin lymphoma (NHL). Rituximab is often used to treat WM and IgM MGUS neuropathies. Biosimilars are FDA approved drugs that have been determined to be interchangeable with the original drug.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate. Screening evaluations including consent, physical exam, and laboratory assessments will be done within 30 days prior to Cycle 1 Day 1. Bone marrow biopsy &aspirate, skin (fat) biopsy, EMG, and CT C/A/P will be done within 90 days prior to Cycle1 Day 1.
* Presence of an IgM monoclonal paraprotein on serum immunofixation electrophoresis
* Diagnosis of IgM MGUS or Waldenstrӧm macroglobulinemia using the criteria from Owen RG, Treon SP, Al-Katib A, Fonseca R, Greipp PR, McMaster ML, et al.Clinicopathological definition of Waldenstrom's macroglobulinemia: consensus panel recommendations from the Second International Workshop on Waldenstrom's Macroglobulinemia. Semin Oncol. 2003. 30(2): 110-5.

  * WM diagnostic criteria

    * IgM monoclonal gammopathy of any concentration
    * Bone marrow infiltration by small lymphocytes showing plasmacytoid/plasma cell differentiation
    * Intertrabecular pattern of bone marrow infiltration
  * Surface IgM+, CD5 +/-, CD10-, CD19+, CD20+, CD22+, CD23-, CD25+, CD27+, FMC7+, CD103-, CD138- immunophenotype* --- Variations from this immunophenotypic profile can occur. However, care should be taken to satisfactorily exclude other lymphoproliferative disorders. This is most relevant in CD5+ cases, for which chronic lymphocytic leukemia and mantle cell lymphoma require specific exclusion before a diagnosis of WM can be made.
* IgM MGUS diagnostic criteria

  * IgM monoclonal gammopathy of any concentration
  * No bone marrow infiltration
* Presence of predominantly sensory neuropathy with predominant demyelinating features on nerve conduction studies.
* Modified Rankin Scale score of ≥1 with progressing symptoms or a score ≥2
* ECOG ≤2
* Age > 18 years
* Participants may not be on any active therapy for other malignancies with the exception of topical therapies for basal cell or squamous cell cancers of the skin
* At the time of screening, participants must have acceptable organ and marrow function as defined below:

  * Absolute neutrophil count≥1,000/uL (no growth factor permitted within previous 7 days)
  * Platelets ≥100,000/uL (no platelet transfusions permitted within previous 7 days); patients may enroll below this threshold if not attributable to IgM MGUS or WM after consultation with Sponsor-Investigator.
  * For participants with platelets <100,000 uL deemed to be attributable to other causes than IgM MGUS or WM, platelets must be ≥50,000 uL (no platelet transfusions permitted)
* Hemoglobin ≥ 10 g/dL (transfusions permitted); patients may enroll below this threshold if not attributable to IgM MGUS or WM after consultation with Sponsor-Investigator.

  -- For participants with hemoglobin <10 g/dL deemed to be attributable to other causes than IgM MGUS or WM, hemoglobin must be ≥7 g/dL(transfusions permitted)
* Total bilirubin < 1.5 x institutional ULN
* AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN
* Estimated GFR ≥30 mL/min
* International normalized ratio (INR) ≤ 2 x ULN and activated partial thromboplastin time (aPTT) ≤ 2 x ULN. Patients with INR and/or aPTT >2 x ULN who have lupus anticoagulant may be enrolled.
* Females of childbearing potential (FCBP) must use highly effective contraception (see Appendix D) or have complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) while participating in the study; and 2) for at least 1 week after last dose of acalabrutinib and 12 months from last dose of rituximab/biosimilar. FCBP must be referred to a qualified provider of contraceptive methods if needed. FCBP must have a negative serum pregnancy test at screening.
* Men must agree to use a latex condom during treatment and for up to 1 week after the last dose of acalabrutinib and 12 months after the last dose of rituximab during sexual contact with a FCBP
* Ability to adhere to the study visit schedule and other protocol requirements
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study:
* Serum IgM ≥4,000 mg/dL
* Waldenstrӧm macroglobulinemia meeting criteria for treatment using consensus panel criteria from the Second International Workshop on WM besides symptomatic peripheral neuropathy.
* Prior exposure to chemotherapy, BTK inhibitors or other therapies used for WM treatment, except steroids, IVIG, or anti-CD20 antibodies that were administered >90 days prior to first dose of study drug
* Concurrent participation in another therapeutic clinical trial.
* Participants with marginal zone lymphoma (MZL), chronic lymphocytic leukemia (CLL), mantle cell lymphoma (MCL), IgM Myeloma or AL amyloidosis are excluded (Diagnosis based on WHO Classification of Tumours of Hematopoietic and Lymphoid Tissues, S.H. Swerdlow, et al., Editors. 2017, IARC)
* Uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP)
* Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months prior to screening
* Prior hypersensitivity, anaphylaxis, or intolerance to rituximab/biosimilar and ofatumumab, or acalabrutinib, including active product or excipient components
* Vaccination with a live vaccine within 4 weeks prior to first dose of rituximab.
* Prior or concurrent active malignancy within the past 2 years, except for curatively treated basal or squamous cell skin cancer, carcinoma in situ of the cervix or breast, or localized prostate cancer.
* Any condition, including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study
* Known history of neuropathy attributed to an etiology other than IgM-mediated neuropathy
* Concurrent administration of medications that are moderate or strong inhibitors or inducers of CYP3A within 7 days prior to first dose of study drug
* Current, ongoing daily use of a proton pump inhibitor. Participants who switch to H2- receptor antagonists or antacids are eligible.
* Participants with chronic liver disease and hepatic impairment meeting Child-Pugh class C
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists
* Peripheral neuropathy symptoms that have been present for >5 years
* Known central nervous system lymphoma
* Active bleeding or history of bleeding diathesis (e.g., congenital von Willebrand's disease or hemophilia)
* History of significant cerebrovascular disease/event, including stroke or intracranial hemorrhage, within 6 months prior to the first dose of study drug
* Major surgery within 4 weeks of first dose of study drug
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Female participants who are pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 1 week of last dose of study drug acalabrutinib, or 12 months of last dose of rituximab/biosimilar.
* Male participants who plan to father a child while enrolled in this study or within 90 days after the last dose of study drug
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening
* New York Heart Association classification III or IV heart failure
* No active Human Immunodeficiency Virus (HIV) infection
* Active infection with Hepatitis B virus (HBV) or viral hepatitis C (HCV) as follows:

  * Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Note: Patients with presence of HBcAb, but absence of HBsAg, are eligible if HBV DNA is undetectable and if they are willing to undergo monitoring for HBV reactivation throughout the study.
  * Patients with presence of HCV antibody are eligible if HCV RNA is undetectable and if they are willing to undergo monitoring for HCV reactivation.
* No significant infection (eg bacterial, viral, or fungal) at study entry
* Inability to swallow pills
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Unwillingness or inability to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall hematologic response rate | baseline to 6 years
  defined as ≥25% reduction in serum IgM) during treatment compared to baseline in patients with IgM mediated symptomatic neuropathy treated with the combination acalabrutinib + rituximab (or biosimilar

SECONDARY OUTCOMES:
Progression Free Survival | Duration of time from start of treatment to time of objective disease progression (including initiation of new therapy or death) up to 6 years
  Time from initiation of Acalabrutinib + rituximab therapy until disease progression (>25% increase in serum IgM and 500 mg/dL absolute increase).
Time to next treatment | Duration of time from start of treatment to next therapy or last follow-up up to 72 months
  Time from initiation of Acalabrutinib + rituximab therapy until initiation of new line of therapy
Overall Survival | Duration of time from start of treatment to time of death or last follow-up up to 72 months
  Time from initiation of therapy until death
Complete Response Rate | Duration of time from start of treatment to last follow-up up to 72 months.
  Proportion of patients with a complete response. Complete response (CR) is defined as having resolution of WM related symptoms, normalization of serum IgM levels with complete disappearance of IgM paraprotein by immunofixation, and resolution of any adenopathy or splenomegaly. A complete response requires reconfirmation demonstrating normal serum IgM levels, and absence of IgM paraprotein by immunofixation by a measurement repeated at least 2 weeks later.
Bone marrow response | Cycle 12, yearly up to 4 years
  Absolute change in bone marrow burden of disease from baseline in patients who have involvement at baseline.
Number of Participants to Treatment Related Adverse Events | Throughout the study and for 30 days after the last dose, up 4 years
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Very Good Partial Response (VGPR): | Duration of time from start of treatment to last follow-up up to 72 months.
  Proportion of patients with a very good partial response (VGPR) defined as >90% reduction in serum IgM levels, or normalization of serum IgM levels with persistent IgM monoclonal spike in SPEP or immunofixation.
Partial Response (PR): | Duration of time from start of treatment to last follow-up up to 72 months.
  Proportion of patients with a Partial response (PR) is defined as achieving a >50% reduction in serum IgM levels.
Minor Response (MR): | Duration of time from start of treatment to last follow-up up to 72 months.
  Proportion of patients with a minor response (MR) is defined 25-49% reduction in serum IgM levels.
Rate of neuropathy response by INCAT-ISS | Cycles 3, 6, 9, 12 (each cycle is 28 days), and then yearly for the duration of the study up to 6 Years
  The proportion of patients with improvement or stability in neuropathy based on INCAT-ISS
Rate of neuropathy response by INCAT disability score | Cycles 3, 6, 9, 12 (each cycle is 28 days), and then yearly for the duration of the study up to 6 Years
  The proportion of patients with improvement or stability in neuropathy based on INCAT disability score
Rate of neuropathy response by MRC distal sum score | Cycles 3, 6, 9, 12 (each cycle is 28 days), and then yearly for the duration of the study up to 6 Years
  The proportion of patients with improvement or stability in neuropathy based on MRC distal sum score
Rate of neuropathy response by 10-meter walk time | Cycles 3, 6, 9, 12 (each cycle is 28 days), and then yearly for the duration of the study up to 6 Years
  The proportion of patients with improvement or stability in neuropathy based on 10-meter walk time changes.
Rate of neuropathy response by 9-hole peg test | Cycles 3, 6, 9, 12 (each cycle is 28 days), and then yearly for the duration of the study up to 6 Years
  The proportion of patients with improvement or stability in neuropathy based on 9-hole peg test.
Rate of neuropathy response by VAS | Cycles 3, 6, 9, 12 (each cycle is 28 days), and then yearly for the duration of the study up to 6 Years
  The proportion of patients with improvement or stability in neuropathy based on Visual Analogue Scale.
Rate of neuropathy response by I-RODS functional score | Cycles 3, 6, 9, 12 (each cycle is 28 days), and then yearly for the duration of the study up to 6 Years
  The proportion of patients with improvement or stability in neuropathy based on I-RODS functional score
Rate of neuropathy response by Rausch built FSS | Cycles 3, 6, 9, 12 (each cycle is 28 days), and then yearly for the duration of the study up to 6 Years
  The proportion of patients with improvement or stability in neuropathy based on Rausch built Fatigue Severity Score
Rate of neuropathy response by IN-QOL tool | Cycles 3, 6, 9, 12 (each cycle is 28 days), and then yearly for the duration of the study up to 6 Years
  The proportion of patients with improvement or stability in neuropathy based on IN-QOL tool

CONTACTS AND LOCATIONS:
Overall Officials: Shayna R. Sarosiek, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Nardin J, Dittus C, Traub R. Clinical and Electrodiagnostic Findings in Anti-myelin-Associated Glycoprotein Antibody Polyneuropathy: A Single Center Review. J Clin Neuromuscul Dis. 2025 Jun 2;26(4):200-205. doi: 10.1097/CND.0000000000000525. PMID 40513035